CLINICAL TRIAL: NCT03275116
Title: The Effect of Twice Daily Aclidinium Bromide/Formoterol Fumarate 340/12 mcg vs. Once Daily Tiotropium 'Respimat' 5mcg on Static and Dynamic Hyperinflation in Patients With COPD During 24 Hours
Brief Title: The Effect of Twice Daily vs. Once Daily Bronchodilation on Hyperinflation in COPD Patients During 24 Hours.
Acronym: BOTH
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Center for Integrated Rehabilitation and Organ Failure Horn (Other); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 59452
Record Dates: First submitted 2016-11-08; First posted 2017-09-07 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Chronic Obstructive Airway Disease
Keywords: Bronchodilation; Hyperinflation; Physical activity; Sleep quality
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity; Sleep Initiation and Maintenance Disorders | interventions — aclidinium bromide; Formoterol Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Twice daily dual bronchodilation (Active Comparator): Twice daily Aclidinium Bromide/Formoterol Fumarate 340/12 mcg during 4 days
  Interventions: Drug: Tiotropium 'Respimat' 5 mcg
- Once daily single bronchodilation (Active Comparator): Once daily Tiotropium 'Respimat' 5 mcg during 4 days
  Interventions: Drug: Aclidinium Bromide/Formoterol Fumarate 340/12 mcg

INTERVENTIONS:
Drug: Tiotropium 'Respimat' 5 mcg — Once daily single bronchodilation
  Other Names: Spiriva 'Respimat'
  Arms: Twice daily dual bronchodilation
Drug: Aclidinium Bromide/Formoterol Fumarate 340/12 mcg — Twice daily dual bronchodilation
  Other Names: Duaklir Genuair
  Arms: Once daily single bronchodilation

SUMMARY:
To study the effect of twice daily dual bronchodilation versus once daily single bronchodilation in patients with chronic obstructive pulmonary disease on 24-hour static and dynamic hyperinflation.

DETAILED DESCRIPTION:
To study the effect of twice daily dual bronchodilation (Aclidinium Bromide/Formoterol Fumarate 340/12 mcg) versus once daily single bronchodilation (Tiotropium 'respimat' 5 mcg) in patients with COPD on 24-hour static and dynamic hyperinflation, spirometry respiratory symptoms and sleep quality.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults (with an equal sex ratio not exceeding 35-65%) aged ≥ 40 years with written informed consent obtained prior to any study-related procedure.
2. Patients entering pulmonary rehabilitation at CIRO.
3. Patients with a diagnosis of moderate to very severe COPD at least 12 months before the screening visit (A post-bronchodilator FEV1 < 80% of the predicted normal value and a post-bronchodilator FEV1/FVC < 0.7 at least 10-15 min after 4 puffs (4 x 100 μg) of salbutamol)
4. Patients with severe static hyperinflation defined as residual volume (body box) > 150 % predicted.
5. Current smokers or ex-smokers with a smoking history of at least 10 pack years [pack-years = (number of cigarettes per day x number of years)/20].
6. MMRC (modified Medical Research Council Dyspnea scale) score ≥ 2.
7. A cooperative attitude and ability to use correctly the inhalers. ICS (inhalation corticosteroids) use is not an exclusion criterion for participation in the study and will be continued during the study. During the study, patients receive fluticasone in an equivalent dose of their own regimen.

The use of neomacrolides and/or leukotriene antagonists is not an exclusion criterion for participation in the study and will be continued in the study, as long as there are no changes in the regiments in the 4 weeks prior to the study. Also, the use of corticosteroid maintenance therapy is allowed, provided that no changes in the regiments took place in the 4 weeks prior to study.

Exclusion Criteria:

1. Pregnant or lactating women and all women physiologically capable of becoming pregnant (i.e. women of childbearing potential)
2. Patients requiring use of the following medications:

   1. A course of systemic steroids longer than 3 days for COPD exacerbation in the 4 weeks prior to screening.
   2. A course of antibiotics for COPD exacerbation longer than 7 days in the 4 weeks prior to screening. NB; maintenance treatment of macrolides is allowed, without any changes in the regimen in the 4 weeks prior to the study.
   3. PDE4 (phosphodiesterase-4) inhibitors in the 4 weeks prior to screening.
   4. Xanthines in the 4 weeks prior to screening.
   5. Use of antibiotics for a lower respiratory tract infection (e.g pneumonia) in the 4 weeks prior to screening.
3. COPD exacerbation requiring prescriptions of systemic corticosteroids and/or antibiotics or hospitalization during the run-in period.
4. Patients treated with non-cardio selective β-blockers in the month preceding the screening visit or during the run-in period. Those patients may enter the study after non-selective β-blockers withdrawal and/or cardio selective β-blockers intake for at least 10 days before the first study day.
5. Patients treated with long-acting antihistamines unless taken at stable regimen at least 2 months prior to screening and to be maintained constant during the study, or if taken as PRN (Pro Re Nata).
6. Patients requiring long term (at least 12 hours daily) oxygen therapy for chronic hypoxemia.
7. Known respiratory disorders other than COPD which may impact the efficacy of the study drug according the investigator's judgment. This can include but is not limited to alpha-1 antitrypsin deficiency, active tuberculosis, a history of asthma, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension and interstitial lung disease.
8. Previous lung surgery or endoscopic lung volume reduction interventions.
9. Patients who have clinically significant cardiovascular condition such as, but not limited to, unstable ischemic heart disease, NYHA Class III/IV left ventricular failure, acute ischemic heart disease in the last year prior to study screening, history of sustained cardiac arrhythmias or sustained and non-sustained cardiac arrhythmias diagnosed in the last 6 months (sustained means lasting more than 30 seconds and or ending only with external action, and or leads to hemodynamic collapse; non-sustained means > 3 beats < 30 seconds, and or ending spontaneously, and or asymptomatic), impulse conduction high degree blocks, patients with Implantable Cardioverter Defribrillator (ICD).
10. Patients with atrial fibrillation (AF):

    1. Paroxysmal Atrial Fibrillation
    2. Persistent: AF episode either lasts longer than 7 days or requires termination by cardioversion, either with drugs or by direct current cardioversion (DCC) within 6 months from screening.
    3. Long standing persistent as defined by continuous atrial fibrillation diagnosed for less than 6 months with or without a rhythm control strategy.
    4. Permanent: for at least 6 months with a resting ventricular rate ≥ 100/min controlled with a rate control strategy (i.e., selective β-blocker, calcium channel blocker, pacemaker placement, digoxin or ablation therapy).
11. An abnormal and clinically significant 12-lead ECG which may impact the safety of the patient according to investigator's judgement. Patients whose electrocardiogram (ECG12 lead) shows QTcF >450 ms for males or QTcF >470 ms for females at screening visit are not eligible (not applicable for patient with pacemaker).
12. Medical diagnosis of narrow-angle glaucoma, prostatic hypertrophy or bladder neck obstruction that in the opinion of the investigator would prevent use of anticholinergic agents.
13. History of hypersensitivity to anticholinergics, β2-agonist or any of the excipients contained in any of the formulations used in the trial which may raise contra-indications or impact the efficacy of the study drug according to the investigator's judgement.
14. Clinically significant laboratory abnormalities indicating a significant or unstable concomitant disease which may impact the efficacy or the safety of the study drug according to investigator's judgement.
15. Patients with hypokalaemia (serum potassium levels <3.5 mEq/L (or 3.5 mmol/L)) or uncontrolled hyperkalaemia according to investigator's judgment.
16. Unstable concurrent disease: e.g. uncontrolled hyperthyroidism, uncontrolled diabetes mellitus or other endocrine disease; significant hepatic impairment; significant renal impairment; uncontrolled gastrointestinal disease (e.g. active peptic ulcer); uncontrolled neurological disease; uncontrolled haematological disease; uncontrolled autoimmune disorders, or other which may impact the efficacy or the safety of the study drug according to investigator's judgment.
17. Patients with any history of malignancy likely to result in significant disability or likely to require significant medical or surgical intervention within the next six months (after V1) or with malignancy for which they are currently undergoing radiation therapy or chemotherapy.
18. History of alcohol abuse and/or substance/drug abuse within 12 months prior to screening visit.
19. Participation in another clinical trial where investigation drug was received less than 8 weeks prior to screening visit.
20. Patients with hypercapnia (≥6.5 kPa) in the arterial blood gas. At screening visit (V1), all exclusion criteria will be checked.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2017-07-07 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Static hyperinflation | 24 hours
  Residual volume (RV) measured by repeated body box measurements

SECONDARY OUTCOMES:
Dynamic hyperinflation | 24 hours
  ∆ICMPT (inspiratory capacity, measured by metronome paced tachypnea)
Airway obstruction | 24 hours
  Measured by FEV1 (forced expiratory capacity in 1 second) by repeated spirometry
Forced vital capacity | 24 hours
  Measured by FVC (forced vital capacity) by repeated spirometry
Inspiratory vital capacity | 24 hours
  Measured by IVC (inspiratory vital capacity) by repeated spirometry
Momentarily symptoms of dyspnea | 24 hours
  Momentarily symptoms of dyspnea during 24 hours will be measured by the BORG scale on dyspnea.
Respiratory symptoms | 4 days
  Dyspnea throughout the week will be measured by the Baseline Dyspnea Index and the Transition Dyspnea Index
Night-time awakenings due to respiratory symptoms | 4 days
  Quality of sleep will be measured using night-time awakening scores, counting the night-time awakenings due to COPD symptoms (wheezing, shortness of breath and coughing). Also a VAS score for sleep quality will be used. A visual score in which patients will assign a number from 0-10 on the question: "How did you sleep the last few days?". In wich 0 is "couldn't be worse" and 10 is "couldn't be better".
Sleep quality | 4 days
  A visual score in which patients will assign a number from 0-10 on the question: "How did you sleep the last few days?". In wich 0 is "couldn't be worse" and 10 is "couldn't be better".
Nighttime physical activity | 4 days
  Measured by an accelerometer, as inverse surrogate for sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: Lowie Vanfleteren, MD, PhD, Principal Investigator — CIRO, centre of expertise for chronic organ failure
Locations (1):
- Ciro, center of expertise in chronic organ failure, Horn, Netherlands